CLINICAL TRIAL: NCT04168944
Title: A Randomized Controlled Study of Lenvatinib Following Liver Transplantation in Patients With High-Risk Hepatocellular Carcinoma
Brief Title: Lenvatinib Following Liver Transplantation in Patients With High-Risk Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2019059
Record Dates: First submitted 2019-11-08; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study were randomly allocated in the lenvatinib group (54 patients) and the control group (54 patients) after stable condition.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- lenvatinib group (Experimental): Participants are given the same anti-rejection therapy as the control group after liver transplantation. 1-2 months after liver transplantation, participants are given lenvatinib with an initial dose of 8 mgor 12 mg orally once a day. The initial dose was 8 mgor 12 mg orally once a day.
  Interventions: Drug: Lenvatinib; Drug: Immunosuppressive regimen
- Placebo group (Placebo Comparator): Immunosuppressive regimen consisting of calcineurin inhibitor, mycophenolate mofetil, sirolimus or ivermus
  Interventions: Drug: Placebo; Drug: Immunosuppressive regimen

INTERVENTIONS:
Drug: Lenvatinib — Patients in the lenvatinib group are given lenvatinib within 1-2 months after operation
  Other Names: E7080
  Arms: lenvatinib group
Drug: Placebo — Sugar pill manufactured to mimic Lenvatinib 10mg tablet
  Arms: Placebo group
Drug: Immunosuppressive regimen — Immunosuppressive regimen consisting of calcineurin inhibitor, mycophenolate mofetil, sirolimus or ivermus

SUMMARY:
The aim of this study is to observe the efficacy and safety of lenvatinib in preventing high-risk recurrence of hepatocellular carcinoma patients after liver transplantation.The cases are from patients with hepatocellular carcinoma who underwent liver transplantation in the liver surgery department of Shanghai Renji Hospital. Patients enrolled in the study were randomly allocated in the lenvatinib group (54 patients) and the control group (54 patients) after stable condition.

DETAILED DESCRIPTION:
The research is an open, randomized, single-center study. Patients with high-risk recurrence of hepatocellular carcinoma who underwent liver transplantation are included according to the criteria of admission. After operation, the regimen of calcineurin inhibitors, mycophenolate mofetil, sirolimus or everolimus with glucocorticoids removed at an early stage are used. Patients enrolled in the study were randomly allocated in the lenvatinib group (54 patients) and the control group (54 patients) after stable condition. Patients in the control group are given supportive treatment and regular follow-up. Patients in the lenvatinib group are given lenvatinib within 1-2 months after operation (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day). The baseline data of patients are collected before allocation. Serum and imaging examination are checked regularly every month to monitor the recurrence of hepatocellular carcinoma and the side effects of lenvatinib. The efficacy and safety of lenvatinib in patients of high-risk hepatocellular carcinoma are observed, and the clinicopathological factors affecting the efficacy of lenvatinib are analyzed. When side effects of lenvatinib occur, the dosage can be reduced according to the patients' condition until discontinuation. When tumor recurrence occurs, a multidisciplinary team will draw up specific treatment plans according to the patients' condition, including surgical resection, interventional therapy, radiofrequency therapy, radiotherapy and targeted therapy (Patients in the control group can add lenvatinib, and patients in the lenvatinib group can decide whether to continue using it according to the patients' condition).

ELIGIBILITY:
Inclusion Criteria:

* Patients at high risk of recurrence of hepatocellular carcinoma after liver transplantation: extended Milan criteria, without vascular invasion (except for microvascular invasion suggested by pathology after operation)

  * Male or female patients aged 18 to 75.

    * ECOG physical condition was 0-2 points.

      * Child-Pugh A grade of liver function.

        * Targeted therapy is acceptable within 1-2 months after liver transplantation. ⑥Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.

          ⑦No history of surgical resection of liver tumors and targeted drug therapy before liver transplantation.

          ⑧Good liver, kidney and bone marrow function: serum albumin > 28g/L, total bilirubin ≤ 3 mg/dL (51.3 umol/l), ALT and AST ≤ 5 times the upper limit of normal range; serum creatinine ≤ 1.5 times the upper limit of normal range; hemoglobin > 90 g/L, neutrophil count (ANC) > 1.5 * 10 ^ 9/L, platelet count > 60 * 10 ^ 9/L; PT-INR < 2.3, or PT within 6 seconds over normal upper limit.

          ⑧For fertile female patients, the serum/urine pregnancy test should be negative within 7 days before treatment.

          ⑨All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.

          ⑩The participants have the capability of oral medication.

          ⑾The participants must sign the consent form.

Exclusion Criteria:

* Life expectancy is less than 3 months

  * The recurrence and metastasis of hepatocellular carcinoma are highly suspected.

    * Patients are with other malignant tumors simultaneously.

      * Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.

        * Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).

          * Preoperative history of severe cardiovascular disease: congestive heart failure > NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.

            * History of HIV infection.

              ⑧Severe clinical active infections (> NCI-CTCAE version 3.0).

              ⑨Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).

              ⑩Patients with kidney diseases requires renal dialysis.

              ⑾Drug abuse, medical symptoms, mental illness or social status that may interfere with participants'participation in research or evaluation of research results.

              ⑿Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.

              ⒀Other anti-angiogenesis therapies, surgery, TACE, local therapy and systemic chemotherapy were given before the treatment after liver transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Tumor free survival rate | 5 years
  The 1, 3, 5-year of tumor free survival rate

SECONDARY OUTCOMES:
Overall survival rate | 5 years
  The 1, 3, 5-year of overall survival rate

OTHER OUTCOMES:
the side effects | 5 years
  The side effects during treatment were recorded. At the same time, patients status will be scored according to ECOG PS score. Acute or subacute toxicity is classified as level of 0-4, 0 as non-response, 1 as mild, 2 as moderate, 3 as severe and 4 as life-threatening. The severity of adverse events was judged, reported and handled according to GCP requirements of clinical trials.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04168944/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT04168944/ICF_001.pdf